CLINICAL TRIAL: NCT05231707
Title: A Couples-focused Intervention for HIV Prevention and Care in South Africa
Brief Title: Simunye: A Couples-focused Intervention for HIV Prevention and Care in South Africa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of California, San Francisco (Other); Human Sciences Research Council (Other Government)
Responsible Party: Principal Investigator, Lynae Darbes, Professor of Nursing, School of Nursing, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00203672
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Couples
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): For couples who are prevalent sero-discordant, this will be a CHTC session. For couples who are prevalent concordant HIV-positive, the first visit will be the first Partner Steps session. For couples in which one or both do not know their sero-status or have not tested for HIV in the past 12 months, the first session will be a CHTC session.
  Interventions: Behavioral: A couples-focused intervention for HIV prevention and care in South Africa
- Attention Matched Control (Active Comparator): Participants in the control group will receive an intervention, with the same number of sessions as couples of the same sero-status in the intervention condition, delivered via one-on-one couples counseling sessions (i.e., one couple with one counselor).
  Interventions: Behavioral: A couples-focused intervention for HIV prevention and care in South Africa

INTERVENTIONS:
Behavioral: A couples-focused intervention for HIV prevention and care in South Africa — From a sample of 272 male-female couples (544 individuals, 272 men and 272 women) recruited from rural KaZulu-Natal, South Africa, couples will be randomized to receive either individual a package of dyadic counseling and testing (intervention arm) or an attention matched control.

SUMMARY:
From a sample of 272 male-female couples (544 individuals, 272 men and 272 women) recruited from rural KaZulu-Natal, South Africa, couples will be randomized to receive either individual a package of dyadic counseling and testing (intervention arm) or an attention matched control. The research examines the impact of a package of dyadic counseling and testing on viral suppression and engagement in HIV care among sero-discordant and concordant positive male-female couples in KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
South Africa remains one of the countries mostly heavily impacted by the HIV epidemic, with an overall estimated adult HIV prevalence of 18% to 30% among female antenatal clinic attendees. There is now substantial evidence that more than 80% of new infections occur within primary male-female partnerships. The high rates of new infections among primary partnerships are attributed to a combination of low levels of HIV testing and a high prevalence of outside sex partners. Recent work by Darbes (MPI), in KwaZulu-Natal (KZN) - the site of the proposed new research - found that among a sample of 330 heterosexual couples, 49% of men and 41% of women had no previous HIV testing history. In 20% of couples, neither partner had ever tested for HIV, despite living in a region with one of the highest adult HIV prevalence globally. Beyond the low levels of HIV testing, recent work also demonstrates significant deficits across the continuum of care in South Africa: recent work by Haber in KZN shows that only 45% of HIV-positive individuals are linked to care, 35% initiate ART, and 33% reach viral suppression. There is increasing evidence of efficacy for couples' focused HIV prevention interventions. Couples HIV Testing and Counseling (CHTC) is a proven strategy to reduce the risk of HIV transmission between partners. However, CHTC focuses only on the first stage of the cascade of HIV care - testing - are there are no interventions that allow couples to pass through the cascade of care together. Using a randomized controlled trial design with 272 couples, we aim to address this gap in HIV prevention and care literature by comparing a package of dyadic focused HIV testing and counseling interventions, against an attention matched control. The proposed RCT will test the efficacy of the dyadic intervention for achieving gains in viral suppression and engagement in HIV care. Heterosexual couples represent a significant yet over- looked risk group in South Africa, and innovative solutions are urgently needed to improve progression across the continuum of HIV care.

ELIGIBILITY:
Inclusion Criteria:

1. both aged between 18-50
2. report being a cis-gender male and a cis-gender female
3. report being in a relationship with each other for at least 6 months
4. are not in a polygamous marriage and 5) report being sexually active with their partner.

Serostatus Inclusion Criteria:

For those individuals who already know that they are HIV-positive, the inclusion criteria will be that they report one of the following conditions:

1. have never initiated ART
2. not currently on ART (but can have been on it before)
3. if already on ART, that they have missed 3 doses of medication in the past 30 days

Exclusion Criteria:

1. Couples in which one or both members report experiencing or perpetrating severe IPV in the prior 6 months
2. Below age 18 or above age 50
3. Report being transgender
4. Report not being a relationship at all or for <6 months
5. Are in a polyamorous marriage
6. Are not sexual active with participating partner

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender only
Enrollment: 544 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Virologic suppression change | Baseline and every 6 months for 24 months
  A blood draw will be conducted to provide a measure of viral load at each visit to look for changes between visits. The outcome will be a binary outcome of detectable versus undetectable viral load.

SECONDARY OUTCOMES:
Behavioral indicators of engagement in HIV care | Baseline and every 6 months for 24 months
  Engagement in care is conceptualized as including linkage to care and retention in HIV care. For HIV-positive partners who report no engagement in HIV care at baseline, linkage to care is defined as attending at least one clinical care appointment, having at least one CD4 test performed, and having at least one viral load test performed within 6 months of the baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Lynae Darbes, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Human Sciences Research Council, Sweetwaters, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No